CLINICAL TRIAL: NCT03256799
Title: An Open Label Study to Investigate the Role of Ivacaftor for the Treatment of Cystic Fibrosis in Combination With Ataluren (PTC124) in Cystic Fibrosis Patients Using Ataluren for Nonsense Mutations
Brief Title: Evaluation of Ivacaftor in Patients Using Ataluren for Nonsense Mutations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Steven M Rowe, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F161208009
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor; ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivacaftor/Ataluren (Experimental)
  Interventions: Drug: Ivacaftor/Ataluren

INTERVENTIONS:
Drug: Ivacaftor/Ataluren — Both drugs were given in combination for 48 week study period

SUMMARY:
The purpose of this study is to explore the combination of Ataluren and ivacaftor as a treatment for patients with a specific cystic fibrosis mutation

DETAILED DESCRIPTION:
In about 10% of patients with CF, the defect in the gene is known as a stop mutation. This mutation truncates the cystic fibrosis transductive regulator (CFTR) protein production by introducing a premature stop in the messenger RNA (mRNA), this type of mutation is known as a stop mutation. Ataluren is a novel, oral drug that promotes this gene to work effectively and readthrough that premature "stop sign". It is hypothesized that ivacaftor may increase the efficacy of Ataluren by activating a specific protein that may not be functioning properly.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of signed and dated informed consent/assent document(s) indicating that the subject (and/or his parent/legal guardian) has been informed of all pertinent aspects of the trial.
2. Age ≥19 years
3. Body weight ≥16 kg
4. Diagnosis of cystic fibrosis and documentation of the presence of a nonsense mutations of the CFTR gene, as determined by historical genotyping
5. Ability to perform a valid, reproducible spirometry with demonstration of a forced expiratory volume in 1second (FEV1) ≥30% of predicted for age, gender, and height.
6. If the subject is sexually active, willingness to abstain from sexual intercourse or employ a barrier or medical method of contraception during the study drug administration
7. Willingness and ability to comply with all study procedures and assessments.
8. Currently receiving Ataluren for nonsense mutations through other clinical trial access.

Exclusion Criteria:

1. Any change (initiation, change in type of drug, dose modification, schedule modification, interruption, discontinuation, or re-initiation) in a chronic treatment/prophylaxis regimen for CF or for CF-related conditions within 2 weeks prior to screening.
2. Evidence of pulmonary exacerbation or acute upper or lower respiratory tract infection (including viral illnesses) within 2 weeks prior to screening.
3. Ongoing immunosuppressive therapy (other than corticosteroids up to 10mg/d equivalent of prednisone)
4. Ongoing warfarin, phenytoin, or tolbutamide therapy.
5. History of solid organ or hematological transplantation.
6. A history of positive hepatitis B surface antigen test, hepatitis C antibody test, or human immunodeficiency
7. Major complications of lung disease (including massive hemoptysis, pneumothorax, or pleural effusion) within 4 weeks prior to screening.
8. Pregnancy or breast-feeding.
9. Current smoker or a smoking history of ≥10 pack-years (number of cigarette packs/day × number of years smoked).
10. Prior or ongoing medical condition (eg, renal failure, alcoholism, drug abuse, psychiatric condition), medical history, physical findings, ECG findings, or laboratory abnormality that, in the investigator's opinion, could adversely affect the safety of the subject, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.

    -

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2018-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Rowe, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: N of 1 trial
Pre-assignment Details: there was no multiple arms in this study and no multiple groups
Groups:
- Ivacaftor/Ataluren: the combination treatment of Ivacaftor/Ataluren were to be given over a 48 week period
Period: Overall Study
Arm/Group | Ivacaftor/Ataluren
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Ivacaftor/Ataluren: Ivacaftor/Ataluren
Arm/Group | Ivacaftor/Ataluren
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Caucasian, non-hispanic
  Participants
    caucasian, non-hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Lung Function
Description: change in lung function as measured by spirometry
Time Frame: Baseline through 48 weeks
Measure: Number; unit: Liters
Groups:
- Ivacaftor/Ataluren: Ivacaftor/Ataluren combination therapy
Arm/Group | Ivacaftor/Ataluren
Number analyzed (Participants) | 1
Liters | 35

ADVERSE EVENTS:
Time Frame: 4 months from March 2017 through July 2017
Description: two pulmonary exacerbations during the N-of-1 trial, both of which occurred following cessation of combination therapy
Arm/Group | Ivacaftor/Ataluren
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivacaftor/Ataluren (N=1)
pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (2) — two pulmonary exacerbations during the N-of-1 trial, both of which occurred following cessation of combination therapy, potentially implicating

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT03256799/Prot_SAP_ICF_000.pdf